CLINICAL TRIAL: NCT00091936
Title: Implementing Anti-Retroviral Therapy in Resource-Constrained Settings: A Randomized Controlled Trial to Assess the Effect of Integrated Tuberculosis and HIV Care on the Incidence of AIDS-Defining Conditions or Mortality in Subjects Co-Infected With Tuberculosis and HIV
Brief Title: Effectiveness of Directly Observed Therapy in Combined HIV and Tuberculosis Treatment in Resource-limited Settings
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CAPRISA START; CAPRISA 001; START; CIPRA
Record Dates: First submitted 2004-09-20; First posted 2004-09-21 (Estimated); Last update posted 2010-03-29 (Estimated); Status verified 2007-01

CONDITIONS: HIV Infections; Tuberculosis
Keywords: Treatment Naive; Directly Observed Therapy; DOT; TB
MeSH Terms: conditions — HIV Infections; Tuberculosis; Directly Observed Therapy | interventions — Didanosine; efavirenz; Lamivudine

INTERVENTIONS:
Drug: Didanosine
Drug: Efavirenz
Drug: Lamivudine
Drug: Standard TB treatment

SUMMARY:
Tuberculosis (TB), a bacterial infection common in HIV infected people, is a major problem in developing countries. The purpose of this study is to test the effectiveness of a combined treatment strategy using directly observed therapy (DOT) for HIV infected patients with TB. Participants will be recruited from resource-poor communities in Durban, South Africa.

DETAILED DESCRIPTION:
TB is the most common serious infectious complication associated with HIV in sub-Saharan Africa and is also the most common cause of death among HIV infected patients in developing countries. Furthermore, TB in an HIV infected person accelerates the progression of HIV disease and hastens death. This study will evaluate a combined TB and antiretroviral treatment (ART) strategy utilizing DOT in HIV infected people coinfected with TB. This study will compare two treatment strategies: TB and HIV medications given concurrently (integrated arm) and TB treatment completed first, followed by HIV treatment (sequential arm).

This study has two parts. The entire study will last 24 months after participants have been randomly assigned to one of two arms. Arm 1 (integrated arm) participants will receive didanosine (ddI), efavirenz (EFV), and lamivudine (3TC) once daily concurrent with standard TB therapy. ART and TB medications will be provided through DOT on weekdays; participants will take their medications without DOT on weekends. Arm 1 participants will also attend four 15- to 20-minute sessions of an adherence study program at study start, Week 2, Month 2, and 1 to 3 weeks prior to the end of TB therapy.

Arm 2 (sequential arm) participants will first receive DOT-provided TB treatment alone. After completion of TB treatment, participants will receive ddI, EFV, and 3TC once daily without DOT.

Study visits in the first part of the study will occur at screening, study start, Weeks 1, 2, and 3, and every month until the end of the first part of the study at Month 12. Study visits will include blood collection, medical and medication history assessment, a physical exam, and pill counts. Patients will be asked to complete an adherence questionnaire at every study visit and a sexual behavior survey and quality of life questionnaire at study start and Month 6.

ELIGIBILITY:
Inclusion Criteria for First Part of Study:

* HIV infected
* TB infected
* Currently receiving standard anti-TB therapy (isoniazid, rifampicin, ethambutol, and pyrazinamide)
* Currently participating in the Prince Cyril Zulu CDC Directly Observed Therapy (DOT) program and receiving treatment daily either there or in the community with a supervised community nurse or trained health worker
* Intending to stay in the area for the duration of the study
* Willing to participate in all follow-up visits
* Willing to use acceptable forms of contraception
* Female participants must be willing to have regular pregnancy tests during ART

Exclusion Criteria for First Part of Study:

* Have had 28 days or more of cumulative ART prior to study entry. Participants who have taken mother-to-child transmission (MTCT) and postexposure prophylaxis (PEP) prevention treatments are not excluded.
* Less than 10 days or greater than 28 days since starting current TB treatment
* Body temperature greater than 38.5 C (101.3 F)
* Rash, nausea, or vomiting of Grade 3 or higher
* Hospitalized or referred for hospitalization for care and treatment of opportunistic infections, TB, or other causes at screening or enrollment
* CD4 count less than 50 cells/microL within 28 days of study entry
* TB meningitis or TB that has spread to the blood and organs other than the lungs
* History of prior TB treatment or previous active TB episode unresponsive to a standard anti-TB regimen
* History of or current AIDS-defining condition as defined by the World Health Organization (WHO)
* History of or current pancreatitis
* Peripheral neuropathy of Grade 2 or higher
* Currently taking certain medications
* Suspected multidrug resistant (MDR) TB
* Any condition that, in the opinion of the investigator, may interfere with the study
* Participation in any other study that may interfere with this study
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 592 (Estimated)
Dates: Start 2009-08

PRIMARY OUTCOMES:
Diagnosis of an AIDS-defining illness
18-month mortality

CONTACTS AND LOCATIONS:
Overall Officials: Salim S. Abdool Karim, MBChB, PhD, Study Chair — University of KwaZulu
Locations (2):
- South Africa (2):
  - King Edward VIII Hospital, KwaKhangela, Durban
  - Prince Cyril Zulu CDC, KwaKhangela, Durban

REFERENCES:
- [Background] Cahn P, Perez H, Ben G, Ochoa C. Tuberculosis and HIV: a partnership against the most vulnerable. J Int Assoc Physicians AIDS Care (Chic). 2003 Jul-Sep;2(3):106-23. doi: 10.1177/154510970300200303. PMID 14556429
- [Background] Corbett EL, Watt CJ, Walker N, Maher D, Williams BG, Raviglione MC, Dye C. The growing burden of tuberculosis: global trends and interactions with the HIV epidemic. Arch Intern Med. 2003 May 12;163(9):1009-21. doi: 10.1001/archinte.163.9.1009. PMID 12742798
- [Background] de Jong BC, Israelski DM, Corbett EL, Small PM. Clinical management of tuberculosis in the context of HIV infection. Annu Rev Med. 2004;55:283-301. doi: 10.1146/annurev.med.55.091902.103753. PMID 14746522
- [Background] Girardi E, Antonucci G, Vanacore P, Palmieri F, Matteelli A, Iemoli E, Carradori S, Salassa B, Pasticci MB, Raviglione MC, Ippolito G; GISTA-SIMIT Study Group. Tuberculosis in HIV-infected persons in the context of wide availability of highly active antiretroviral therapy. Eur Respir J. 2004 Jul;24(1):11-7. doi: 10.1183/09031936.04.00109303. PMID 15293599
- [Background] Girardi E, Goletti D, Antonucci G, Ippolito G. Tuberculosis and HIV: a deadly interaction. J Biol Regul Homeost Agents. 2001 Jul-Sep;15(3):218-23. PMID 11693427
- [Derived] Gengiah TN, Holford NH, Botha JH, Gray AL, Naidoo K, Abdool Karim SS. The influence of tuberculosis treatment on efavirenz clearance in patients co-infected with HIV and tuberculosis. Eur J Clin Pharmacol. 2012 May;68(5):689-95. doi: 10.1007/s00228-011-1166-5. Epub 2011 Nov 23. PMID 22108776